CLINICAL TRIAL: NCT04435704
Title: Validate a Pharmacodynamic Model of Oxytocin for Peripheral Analgesic Effects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not initiated. No subjects enrolled.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00066138
Record Dates: First submitted 2020-06-04; First posted 2020-06-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Oxytocin will be administered by intravenous infusion at increasing and decreasing rates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oxytocin (Experimental): Oxytocin will be administered at increasing and decreasing rates
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Intravenous Oxytocin
  Other Names: Pitocin

SUMMARY:
The goal of this study is to validate the pharmacodynamic model for pain relief from oxytocin at a peripheral site by intravenous infusion targeted at different levels of the drug.

In this study healthy volunteers and people with knee arthritis so severe that they may need joint replacement are recruited for a one day study. Each study participant will have an intravenous(IV) catheter placed. After placement of the IV catheter oxytocin will be given by IV infusion in varying amounts. The study team will perform some tests to evaluate how oxytocin changes perceptions on the skin. The study team will study a painful perception by placing a probe on the skin and heating it to 113 degrees Fahrenheit for 5 minutes. Each study participant will score any pain that is experienced on a 0 to 10 scale.

DETAILED DESCRIPTION:
This is an unblinded Pharmacokinetic/Pharmacodynamic (PK/PD) study in which oxytocin is infused in increasing steps to different levels up and down in a set manner and the PD effect of pain relief from each level of oxytocin determined. All study participants will receive the same treatment and will not be blinded to the experimental plan, although particpants will not be informed when oxytocin levels are changing.

In this study healthy people or those with knee arthritis so severe that they may need joint replacement are recruited for a one day study. Participants will come to the Clinical Research Unit (CRU) and one intravenous catheter (IV) will be inserted in the forearm for oxytocin infusion. In this study, the oxytocin rate will be changed every 15 minutes for 7 times. Oxytocin will be infused by IV route and 5-min heat pain tests obtained, but instead of giving oxytocin at a constant rate, the rate will be adjusted every 15 minutes to aim to get the right amount at the effect site to reduce pain by 10% of the maximum, then 30%, then 70%, then 90%, then back down to 70%, 30%, and 10%. At the end of each of these 7 15-min infusions participants will be tested for pain with heat and the study team will compare how effective the calculations for the effect site are to control the amount of pain relief obtained at each level.

This information will be analyzed by another group at Stanford University in the PK/PD Core part of this application. Mathematics will be used to calculate how quickly oxytocin moves from the blood to where it reduces pain (Part 1) and to test the accuracy of these calculations (Part 2).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3.
3. For healthy volunteers, normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication. For knee arthritis subjects, normal blood pressure or, for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Verbal pain after heating the skin to 45 degrees Celsius | Baseline at time of infusion
  Prior to the initiation of the oxytocin infusion, the skin will be heated to 45 degrees Celsius for 5 minutes and pain will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Verbal pain after heating the skin to 45 degrees Celsius | 9 minutes after baseline
  10% dose escalation. The skin will be heated to 45 degrees Celsius for 5 minutes and pain will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Verbal pain after heating the skin to 45 degrees Celsius | 24 minutes after baseline
  30% dose escalation. The skin will be heated to 45 degrees Celsius for 5 minutes and pain will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Verbal pain after heating the skin to 45 degrees Celsius | 54 minutes after baseline
  70% dose escalation. The skin will be heated to 45 degrees Celsius for 5 minutes and pain will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Verbal pain after heating the skin to 45 degrees Celsius | 69 minutes after baseline
  90% dose escalation. The skin will be heated to 45 degrees Celsius for 5 minutes and pain will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Verbal pain after heating the skin to 45 degrees Celsius | 84 minutes after baseline
  70% dose de-escalation. The skin will be heated to 45 degrees Celsius for 5 minutes and pain will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Verbal pain after heating the skin to 45 degrees Celsius | 99 minutes after baseline
  30% dose de-escalation. The skin will be heated to 45 degrees Celsius for 5 minutes and pain will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Verbal pain after heating the skin to 45 degrees Celsius | 114 minutes after baseline
  10% dose de-escalation. The skin will be heated to 45 degrees Celsius for 5 minutes and pain will be determined, pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No